CLINICAL TRIAL: NCT01580852
Title: The Effects of Immersion in Dead Sea Water on Glucose Levels in Type 2 Diabetes Mellitus Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Victor Novack (Other)
Responsible Party: Sponsor-Investigator, Victor Novack, Sub Investigator, Soroka University Medical Center
Organization: Soroka University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: sor008412clit
Record Dates: First submitted 2012-04-16; First posted 2012-04-19 (Estimated); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Aquatic Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dead Sea Water (Active Comparator)
  Interventions: Procedure: Dead Sea water
- Pool Water (Sham Comparator)
  Interventions: Procedure: Pool water

INTERVENTIONS:
Procedure: Dead Sea water — Subjects will immerse in mineral (dead sea) waters for twenty minutes twice daily for a period of 10 days
  Arms: Dead Sea Water
Procedure: Pool water — Subjects will immerse in sweet(pool)waters for twenty minutes twice daily for a period of 10 days
  Arms: Pool Water

SUMMARY:
BACKGROUND: Bathing in sweet or mineral water can induce significant physiological changes in several body systems including the endocrine system. To date, there have only been a small number of reports that balneology can reduce blood sugar Levels in patients with type 2 diabetes mellitus (DM].

OBJECTIVE: To compare the effects of a immersion in sweet or mineral water on blood glucose levels in patients with type 2 DM.

METHODS: Forty patients with type 2 DM will immerse in either sweet or mineral water twice daily. In both cases the water will be warmed to a temperature of 35 degrees C and the bath continue for 20 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Uncontrolled type 2 diabetes mellitus patients(HbA1c levels between 7.5-10)
* Ages 18-65
* Signed Informed Consent

Exclusion Criteria:

* Peripheral neuropathy
* Diabetic ulcers or damaged skin
* PVD
* Diabetes diagnosis for over 20 years
* Orthostatic Hypotension

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Glucose Levels | participants will be followed for the duration of hotel stay, an expected average of 5 days

SECONDARY OUTCOMES:
HbA1c levels | three months afer intervention

CONTACTS AND LOCATIONS:
Overall Officials: Idit Liberty, MD, Principal Investigator — Soroka University Medical Center
Locations (1):
- Soroka University Medical Cetner, Beersheba, Israel